CLINICAL TRIAL: NCT01416051
Title: Efficacy of Olibra: A 12 Week Randomized Controlled Trial, and Review of Prior Studies
Brief Title: Efficacy of Olibra: A 12 Week Controlled Trial
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: GNC (Unknown)
Responsible Party: Principal Investigator, Frank Greenway, Principal Investigator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PBRC 25001
Record Dates: First submitted 2011-08-11; First posted 2011-08-12 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test (Active Comparator): Subjects consumed a vegetable oil emulsion in yogurt at a food intake test and were asked to consume the product twice daily for 12 weeks.
  Interventions: Dietary Supplement: Olibra
- Control Group (Placebo Comparator): Subjects were given a placebo of milk fat in yogurt at food intake tests and asked to consume the placebo twice daily for 12 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Olibra — Fractionated palm oil and fractionated oat oil in the proportion of 95:5
  Other Names: Fabuless
  Arms: Test
Other: Placebo — 100% milk fat
  Arms: Control Group

SUMMARY:
Today's obesogenic environment, favors behavioral choices that lead to an excess of energy intake over expenditure, and consequently weight gain. Intervention strategies that harness the body's own appetite and satiety regulating signals could provide an effective means of countering excessive energy intake. The purpose of this study was to investigate whether a vegetable oil emulsion (Olibra) would result in weight loss that was associated with a reduction in food intake.

DETAILED DESCRIPTION:
71 healthy subjects were enrolled (60 females, 11 males; Age: 18 - 60 years, BMI 25 - 40 kg/m2) in a two-phased, randomized, placebo-controlled, double-blind, parallel trial. During a 12-week period, Olibra was compared with a placebo (milk fat). Food intake testing was conducted on three days and anthropometric data was collected on 7 days. Key outcome measures were, body weight, body composition, energy intake, and appetite ratings.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects of both sexes 18 - 60 years of age
* body mass index (BMI) between 25 and 40 kg/m2, inclusive

Exclusion Criteria:

* (1) participation in another clinical trial or receipt of an investigational product 30 days prior to enrollment
* (2) a dietary restraint score of > 13
* (3) weight loss of 4.5 kg or more in the preceding three months
* (4) use of tobacco products, nicotine gum or nicotine patch
* (5) a medical condition or taking regular medication except oral contraceptives and hormone replacement therapy
* (6) use of a nutritional product or dietary supplement or program which might interfere with the conduct of the study or place the subject at risk
* (7) history of alcohol or other drug abuse in the preceding one year
* (8) pregnancy, lactation, post-partum less than six months, planning a pregnancy during the study or not using an acceptable method of contraception
* (9) fasting blood sugar ≥ 126 mg/dl
* (10) known allergy or sensitivity to any ingredient in the supplement
* (11) clinically significant deviations in normal laboratory values
* (12) irregular meal-times, and
* (13) unwilling to eat yogurt at test meals.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2005-01; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Body weight | 12 weeks
  Treatment to determine if test product causes weight loss

SECONDARY OUTCOMES:
Body composition | 12 weeks
  To determine if treatment causes a reduction in body fat mass
Food intake | 4 weeks
  To determine if treatment results in a reduction in food intake

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Derived] Rebello CJ, Martin CK, Johnson WD, O'Neil CE, Greenway FL. Efficacy of Olibra: a 12-week randomized controlled trial and a review of earlier studies. J Diabetes Sci Technol. 2012 May 1;6(3):695-708. doi: 10.1177/193229681200600326. PMID 22768902